CLINICAL TRIAL: NCT07246382
Title: Evaluation of A Customizable Antibiotic Stewardship Program Based on a Comprehensive Assessment of Organizations and Health Professionals' Attitudes, and Tailored to French Nursing Homes' Needs
Brief Title: Evaluation of a Customizable Antibiotic Stewardship Program Tailored to French Nursing Homes
Acronym: ORANEAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lorraine (Other)
Collaborators: Sciences Po, Centre de Sociologie des Organisations (CSO), CNRS, Paris, France. (Unknown); Inserm U1219, Bordeaux Population Health Research Center, Bordeaux, France. (Unknown); Centre Régional en Antibiothérapie (CRAtb) Grand Est, Nancy, France. (Unknown); Centre Régional en Antibiothérapie (CRAtb) Pays de la Loire, Nantes, France. (Unknown); National Research Agency, France (Other); Centre d'appui pour la Prévention des Infections Associées aux Soins (CPias) Pays de la Loire, Nantes, France. (Unknown); Centre d'appui pour la Prévention des Infections Associées aux Soins (CPias) Grand Est, Nancy, France. (Unknown)
Responsible Party: Principal Investigator, Nelly Agriner, Professor, University of Lorraine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ANR-20-PAMR-0008; 21-841 (Other: CEEI IRB00003888, IORG0003254); 2021/170 (Other: French Data Protection Authority)
Record Dates: First submitted 2025-08-22; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Antibacterial Agents
Keywords: Antimicrobial Stewardship; Nursing Homes

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial with two parallel arms (ORANEAT program vs. no specific intervention); the cluster being the nursing home.
Who Masked: Outcomes Assessor
Masking Description: The statisticians responsible for analyzing data on antibiotic use (using data from the Health Insurance reimbursement database, Système national des données de santé)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Nursing homes in the experimental group will receive the ORANEAT antibiotic stewardship program.
  Interventions: Other: The ORANEAT program
- Control group (No Intervention): Nursing homes in the control group will not receive the ORANEAT antibiotic stewardship program ("usual care").

INTERVENTIONS:
Other: The ORANEAT program — The ORANEAT multifaceted customizable antibiotic stewardship program includes (i) a contextual diagnostic regarding AMS in the targeted NH; (ii) based on the results of the contextual diagnostic, a bundle of tools selected from an AMS-toolkit including actions and tools suited to French NH setting and covering the main CDC domains of AMS in NHs; and (iii) implementation support relying on French structures involved in tackling AMR (i.e., CRAtb and CPias).
  Arms: Experimental group

SUMMARY:
To tackle antimicrobial resistance (AMR), i.e., one of the top 10 global health threats, antimicrobial stewardship (AMS) programs, i.e., coherent sets of actions promoting responsible use of antimicrobials, have been developed. Despite growing evidence about their effectiveness, their implementation remains suboptimal. Qualifying as complex interventions, these programs are prone to interactions with context, potentially compromising their successful transfer to other settings. AMR remains critical in French nursing homes (NHs). AMS programs have proven effective in reducing antimicrobial resistance in hospitals and in NHs. However, the evidence is inconsistent across studies in NHs and mostly based on North American and North European AMS programs and studies, raising concerns about transferability that might occur while implementing such AMS programs in French NHs. For instance, health systems and NH funding and organization vary considerably across countries, resulting in potential key determinants driving antibiotic use in such facilities in some countries that might remain untargeted by AMS programs developed in other countries. In addition, inconsistent effectiveness of AMS programs in NHs might also result from implementation issues, raising concerns about the strategies used to implement such programs. Based on extensive logic models linking psychosocial and organizational determinants driving antibiotic use in NHs of diverse countries, we developed and pilot-tested a customizable AMS program (i.e., the ORANEAT program) suited to French NHs, including three major components: (i) a contextual diagnostic regarding AMS in the targeted NH; (ii) based on the results of the contextual diagnostic, a bundle of tools selected from an AMS-toolkit including actions and tools suited to French NH setting; and (iii) implementation support relying on French structures involved in tackling AMR (i.e., CRAtb and CPias).

This study aims to assess the effectiveness, the sustainability, the implementation, and the transferability of the ORANEAT program in French NHs, using a mixed-method approach (quantitative and qualitative data). A cluster randomized controlled trial with two arms (ORANEAT program vs. no specific intervention) will be conducted; the cluster being the NH. The primary outcome to measure the effectiveness is total antibiotic use expressed in defined daily doses/1000 resident-days/month.

ELIGIBILITY:
Nursing homes

Inclusion criteria:

• Nursing home located in one of the geographical areas participating in the study in two French regions (i.e., geographical areas covered by experts in antibiotic stewardship and/or in infection prevention and control who agreed to participate in the study)

Exclusion criteria:

* Nursing home with a pharmacy for internal use
* Participation to the pilot study
* Data from the Health Insurance reimbursement database (Système national des données de santé) not available on the study period
* Refusal of the nursing director to participate in the study (for Arm 1 only)

Residents (Outcomes 1 to 4 and outcome 12)

Inclusion criteria:

• Resident aged 18 or more who had lived in one of the participating nursing homes during the study period.

Exclusion criteria:

/

Healthcare professionals (Outcomes 11, 13 and 15)

Inclusion criteria:

• Healthcare professionals aged 18 or more working in one of the participating nursing homes from Arm 1 (including healthcare professionals who provide services to or collaborate with the nursing home even if they are not on-site, e.g., private general practitioners, community pharmacists, microbiologists, and professionals responsible for the implementation support).

Exclusion criteria:

• Refusal to complete the self-administered questionnaires or to participate in qualitative investigations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Total antibiotic use (DDD) | 12 months
  Total antibiotic use expressed in Defined Daily Doses (DDD)/1000 resident-days/month.
  Measured using data from the Health Insurance reimbursement database.
Total antibiotic use (Number of prescriptions) | 12 months
  As part of a sensibility analysis:
  Total antibiotic use expressed in number of prescriptions/1000 resident-days/month.
  Measured using data from the Health Insurance reimbursement database.

SECONDARY OUTCOMES:
Safety of the intervention | 12 months
  Number of hospital admissions/1000 resident-days and number of deaths/1000 resident-days among nusing home residents.
  Measured using data from the Health Insurance reimbursement database.
Sustainability of the effectiveness | 24 months
  Total antibiotic use expressed in Defined Daily Doses (DDD)/1000 resident-days/month.
  As part of a sensitivity analysis: Total antibiotic use expressed in number of prescriptions/1000 resident-days/month.
  Measured using data from the Health Insurance reimbursement database.

OTHER OUTCOMES:
Context of the intervention - Nursing homes' characteristics | At inclusion
  Nursing homes' staff resources (number of coordinating physicians, nurses, assistant nurses and general practitioners).
  Measured using data collected by the research team through ad hoc standardized activity reports.
Adoption of the intervention | 12 months
  Number of nursing homes included / number of nursing homes invited to participate in the intervention group * 100, by stratum.
  Measured using data collected by the research team through ad hoc standardized activity reports.
Reach of the target population | Through the end of the intervention, an average of 12 months
  Number of copies provided to the nursing home, for each tool (initial number of copies and additional copies requested by the nursing home).
  Measured using data collected by the research team through ad hoc standardized activity reports.
Fidelity of the intervention | Through the end of the intervention, an average of 12 months
  Number of tools used / number of tools included in the bundle of tools, for each bundle.
  Measured using data collected by the by the research team through ad hoc standardized activity reports.
Dose of intervention | Through the end of the intervention, an average of 12 months
  Number of tools used for each target population. Measured using data collected by the by the research team through ad hoc standardized activity reports.
Adaptation of the intervention | Through the end of the intervention, an average of 12 months
  Number of tools withdrawn from the bundle of tools or modified (in form and/or content) or added / number of tools initially proposed (for each bundle of tools and overall).
  Measured using data collected by the by the research team through ad hoc standardized activity reports.
Users' experiences of the intervention | 12 months
  Users' experiences with the ORANEAT program assessed among coordinating physicians/nurses, nurses, assistant nurses and general practitioners using a questionnaire UREMs (User Reported Experience Measures) adapted from PREMs (Patient Reported Experience Measures) developed by the research team. This questionnaire was designed to measure the users reported experience of the intervention. A score ranging from 0 to 100 will be calculated; higher score means better experience.
Sustainability of the intervention | 12 months
  Sustainability of the ORANEAT program assessed among coordinating physicians/nurses, nurses, assistant nurses and general practitioners using the NoMAD questionnaire (questionnaire based on the normalization process theory [NPT], measuring the normalization of complex healthcare interventions - Finch et al. 2018 - doi: 10.1186/s12874-018-0591-x). The NoMAD questionnaire includes three general items on the intervention answered on an 11-point Likert scale ranging from 0 to 10, and 20 items representing the four key constructs of NPT: coherence (4 items), cognitive participation (4 items), collective action (7 items), and reflexive monitoring (5 items) answered on a 5-point Likert scale ranging from strongly agree to strongly disagree. Mean scale scores will be calculated for each NoMAD construct as well as for the overall scale (20 items); higher scores mean higher degree of normalization.
Mechanisms of impact of the intervention - appropriateness of antibiotic prescriptions | 12 months
  Proxy indicators reflecting the appropriateness of antibiotic use in nursing homes (Asquier-Khati et al. 2023, doi:10.1093/jacamr/dlad037). These proxy indicators assess the appropriateness of prescriptions for urinary tract infections, seasonal variations in prescriptions, repeated prescriptions of fluoroquinolones, cephalosporins' route of administration, duration of treatment, rate of second-line antibiotics, and co-prescriptions with non-steroidal anti-inflammatory drugs.
Mechanisms of impact of the intervention - prescriptions of urine cultures | 12 months
  Number of urine cultures prescribed/1000 resident-days/month. Measured using data from the Health Insurance reimbursement database.
Mechanisms of impact of the intervention - nursing home professionals' knowledge, attitudes, practices and motivation | At inclusion, 6 and 12 months
  Nursing home professionals' (coordinating physicians/nurses, nurses, assistant nurses and general practitioners) knowledge, attitudes, practices and motivation towards AMS. For each component (knowledge, attitudes, practices and motivation), a score ranging from 0 to 100 will be calculated; higher scores means more favorable position towards AMS.
  Data collected through the questionnaires of the contextual diagnostic.
Costs of the intervention | Through the end of the intervention, an average of 12 months
  Cost associated with the work provided by the professionals responsible for the implementation support, with printing and sending the ORANEAT program tools to the nursing homes, etc.
  Measured using data collected by the by the research team through ad hoc standardized activity reports.
Context, mechanisms of impact, sustainability, implementation, and transferability of the intervention | Through the end of the intervention, an average of 12 months
  Observations, semi-structured interviews, focus groups with professionals involved in the implementation of the ORANEAT program (coordinating physicians/nurses, nurses, assistant nurses, general practitioners, professionals responsible for the implementation support…).

CONTACTS AND LOCATIONS:
Overall Officials: Nelly AGRINIER, Professor, Principal Investigator — Université de Lorraine, Inserm, INSPIIRE, F-54000 Nancy, France; CHRU-Nancy, Inserm, Université de Lorraine, CIC, Epidémiologie clinique, Nancy, France

IPD SHARING:
Plan to Share IPD: No
IPD Sharing Plan Description: N/A

REFERENCES:
- [Result] Gonthier D, Ricci L, Buzzi M, Birgand G, Kivits J, Agrinier N. Exploration of interprofessional collaboration for the diagnosis of infections and antibiotic prescription in nursing homes using multiple case study observational research. JAC Antimicrob Resist. 2025 Jan 13;7(1):dlae205. doi: 10.1093/jacamr/dlae205. eCollection 2025 Feb. PMID 39807109
- [Result] Bocquier A, Erkilic B, Babinet M, Pulcini C, Agrinier N; ORANEAT Study Group. Resident-, prescriber-, and facility-level factors associated with antibiotic use in long-term care facilities: a systematic review of quantitative studies. Antimicrob Resist Infect Control. 2024 Mar 6;13(1):29. doi: 10.1186/s13756-024-01385-6. PMID 38448955
- [Result] Conlin M, Hamard M, Agrinier N, Birgand G; ORANEAT co-investigators. Assessment of implementation strategies adopted for antimicrobial stewardship interventions in long-term care facilities: a systematic review. Clin Microbiol Infect. 2024 Apr;30(4):431-444. doi: 10.1016/j.cmi.2023.12.020. Epub 2023 Dec 22. PMID 38141820